CLINICAL TRIAL: NCT04484532
Title: Evaluation of Antibody Response to High-Dose Seasonal Influenza Vaccination in Patients With Myeloid Malignancy Receiving Chemotherapy
Brief Title: Evaluation of Antibody Response to High-Dose Seasonal Influenza Vaccination in Patients With Myeloid Malignancy Receiving Chemotherapy and Healthy Volunteers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: I 54017; NCI-2017-02157 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 54017 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2020-07-20; First posted 2020-07-23 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Influenza Vaccines; fluarix; FluBlok; FluLaval; Fluzone High-Dose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Supportive Care (trivalent influenza vaccine) (Experimental): Within 14 days of baseline influenza titer, patients receive trivalent influenza vaccine IM on day 0 (patients in cohorts 1 and 5 receive the vaccine at any time, patients in cohorts 2 and 3 receive the vaccine between days 14-25 of hypomethylating agent therapy course, and patients in cohort 4 receive the vaccine between days 21-365 from onset of cytotoxic chemotherapy). Patients then undergo titer assessment at days 25-90 and days 115-185.
  Interventions: Biological: Trivalent Influenza Vaccine

INTERVENTIONS:
Biological: Trivalent Influenza Vaccine — Given IM
  Other Names: Agriflu; Flu prevention; Flu prophylaxis; Flu shot; Flu vaccination; Fluarix; Flublok; FluLaval; Flushield; Fluvirin; Fluzone High-dose (HD); Influenza Vaccine; Influenza Virus Vaccine, Trivalent, Types A and B; Trivalent Influenza Vaccine (TIV)

SUMMARY:
This pilot research trial studies the antibody response to high-dose seasonal influenza vaccination in patients with myeloid malignancy receiving chemotherapy and healthy volunteers. Evaluating antibody response to high-dose seasonal influenza vaccine may serve as a basis for vaccine recommendations in patients with myeloid malignancies and provide insights into the status of the immune system in these patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To investigate the antibody response to influenza vaccination in patients with acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS) receiving hypomethylating agents (decitabine or azacytidine) compared to normal healthy controls and those patients with similar disorders receiving cytarabine containing intensive chemotherapy or best supportive care.

II. To collect and store blood samples at different time points (prior to and after vaccination) for assessment of influenza specific T-cell subsets using tetramers by flow cytometry.

OUTLINE:

Within 14 days of baseline influenza titer, patients receive trivalent influenza vaccine intramuscularly (IM) on day 0 (patients in cohorts 1 and 5 receive the vaccine at any time, patients in cohorts 2 and 3 receive the vaccine between days 14-25 of hypomethylating agent therapy course, and patients in cohort 4 receive the vaccine between days 21-365 from onset of cytotoxic chemotherapy). Patients then undergo titer assessment at days 25-90 and days 115-185.

ELIGIBILITY:
Inclusion Criteria:

* Subject or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to undergoing any investigational biospecimen (blood) collection procedure
* Willing to undergo seasonal influenza vaccination with Fluzone high dose at Roswell Park Cancer Institute within 2 weeks of enrollment of this study
* Estimated survival of 8 weeks or more following enrollment on the study

Exclusion Criteria:

* Uncontrolled intercurrent illness including, but not limited to, ongoing or active influenza infection or influenza-like-illness
* Women who are attempting pregnancy or known to be pregnant by clinical history or nursing female subjects
* Unwilling or unable to follow protocol requirements
* Use of prednisone > 10 mg/day (or its equivalent for other steroids) for > 2 weeks immediately prior to receiving seasonal influenza vaccination
* Received dose of seasonal influenza vaccination prior to enrollment
* Participation at the time of study enrollment in another clinical trial investigating immunotherapeutic agents (like anti-PD1 or anti-PDL1 or anti-CTLA4 antibodies or vaccines); concurrent participation in an observational/non-interventional study or an interventional study investigating tyrosine kinase inhibitor or other targeted agents use is acceptable
* Inability to receive seasonal influenza vaccine due to prior hypersensitivity to eggs, chicken proteins, or any of the vaccine components
* History of a life-threatening reaction to influenza vaccination or to a vaccine containing similar substances
* Personal history of Guillain-Barre syndrome
* Any condition which in the investigator's opinion deems the subject an unsuitable candidate to receive annual influenza vaccination or may potentially affect the response to influenza vaccination
* Adults unable to consent, individuals who are not yet adults (infants, children, and teenagers), women who are known to be pregnant, attempting pregnancy, or nursing women, and prisoners will be excluded from the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2022-06-07 (Actual)

PRIMARY OUTCOMES:
Antibody response (by microneutralization assay) to influenza vaccination | Up to 4-6 months post-vaccination
  The geometric mean (GMT) and standard deviation of antibody titers will be calculated by cohort at the baseline assessment and 1-3 months post vaccination time points. Antibody response is assessed using the outcome measures: seroprotection, seroconversion, and GMT. Seroprotection is defined as an hemagglutination inhibition (HAI) titer >= 1:40 of each individual influenza antigen. Seroconversion is defined as >= 4-fold increase in post-vaccination titer of each individual influenza antigen. The seroprotection and seroconversion rates will be reported by age strata, cohort, and time-point (1-3 months and 4-6 months post vaccination) using 95% confidence intervals obtained using Jeffrey's prior method. The GMT at each time-point will be compared using one-sided permutation T-tests about the log-transformed data. The GMT ratio (GMTR) between 1-3 months post vaccination and baseline will also be calculated and reported by cohort using a 95% confidence interval.

SECONDARY OUTCOMES:
T-cell subset population assessed using flow cytometry | Up to 4-6 months post-vaccination
  T-cell subset populations will be correlated with antibody responses to influenza vaccination. Blood samples will be collected and stored at different time-points for assessment of T-cell response to influenza vaccination using influenza specific tetramer staining by flow cytometry. The seroprotection and seroconversion rates will be reported by cohort and time-point (1-3 months and 4-6 months post vaccination) using 95% confidence intervals obtained using Jeffrey's prior method. The rates will be compared between the lenalidomide and healthy control cohorts using one-sided Barnard's tests. The GMTR between 1-3 months post vaccination and baseline will also be calculated and reported by cohort using a 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Griffiths, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States